CLINICAL TRIAL: NCT03495102
Title: A Randomized, Double-Blind, Parallel Arm Study of the Efficacy and Safety of Investigational Dulaglutide Doses When Added to Metformin in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of the Efficacy and Safety of Dulaglutide (LY2189265) in Participants With Type 2 Diabetes
Acronym: AWARD-11
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16877; H9X-MC-GBGL (Other: Eli Lilly and Company); 2017-003490-33 (EudraCT Number)
Record Dates: First submitted 2018-04-02; First posted 2018-04-11 (Actual); Results first posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2019-12-15

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dulaglutide 1.5 mg (Active Comparator): Dulaglutide 1.5 mg administered subcutaneously (SC) once a week.
  Interventions: Drug: Dulaglutide
- Dulaglutide 3 mg (Experimental): Dulaglutide 3 mg administered SC once a week.
  Interventions: Drug: Dulaglutide
- Dulaglutide 4.5 mg (Experimental): Dulaglutide 4.5 mg administered SC once a week.
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of investigational doses of once weekly dulaglutide when added to metformin in participants with type 2 diabetes with inadequate blood sugar control.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (T2DM) for at least 6 months
* Have been treated with stable metformin dose for at least 3 months
* Have HbA1c ≥7.5% and ≤11.0% at study entry
* Have body mass index (BMI) ≥25 kilograms per meter squared (kg/m^2)

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have used any glucagon-like peptide-1 receptor agonist (GLP-1 RA) or insulin, not including prior short term insulin use (≤14 days)
* Have been taking any other medicine for diabetes (other than metformin) during the last 3 months
* Have used in the last 3 months (or plan to use) prescription weight loss medications
* Have disorders associated with slowed emptying of the stomach contents, or have had any stomach surgeries for the purpose of weight loss
* Current participation in or intent to begin during the study an organized diet and/or exercise weight reduction program (other than the lifestyle and dietary measures for diabetes)
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease (NAFLD), or alanine transaminase (ALT) level >2.5 times the upper limit of the reference range, as determined by the central laboratory at study entry; participants with NAFLD are eligible for participation in this trial
* Had chronic or acute pancreatitis any time prior to study entry
* Have had a heart attack or stroke in the past 2 months, or have heart failure that significantly limits their physical activity
* Estimated glomerular filtration rate (eGFR) <30 milliliters/minute/1.73m^2 (or lower than the country-specific threshold for discontinuing metformin therapy per local label), calculated by the Chronic Kidney Disease-Epidemiology (CKD-EPI) equation, as determined by the central laboratory at study entry and confirmed at lead-in
* Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2
* Have proliferative retinopathy or maculopathy requiring acute treatment according to the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1842 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (208):
- United States (72):
  - Synexus- Chandler, Chandler, Arizona
  - Synexus/Central Arizona Medical Associates, PC, Mesa, Arizona
  - Central Phoenix Med Clinic LLC, Phoenix, Arizona
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Valley Research, Fresno, California
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Pacific Research Partners, LLC, Oakland, California
  - National Research Institute, Panorama City, California
  - Sierra Clinical Research, Roseville, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Care Access Research, Santa Clarita, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - Diablo Clinical Research, Walnut Creek, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - ALL Medical Research, LLC, Cooper City, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - Urban Family Practice Associates, PC, Marietta, Georgia
  - In-Quest Medical Research, LLC- Peachtree Corners, Peachtree Corners, Georgia
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - East West Medical Institute, Honolulu, Hawaii
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - Saltzer Medical Group. P.A., Nampa, Idaho
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Synexus/Clinical Research Advantage, Evansville, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Iderc, P.L.C., West Des Moines, Iowa
  - InterMed, PA, Portland, Maine
  - MedStar Health Research Institute, Hyattsville, Maryland
  - NECCR PrimaCare Research, LLC, Fall River, Massachusetts
  - Aa Mrc Llc, Flint, Michigan
  - Troy Internal Medicine, PC, Troy, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Montana Health Research, Billings, Montana
  - Glacier View Research Institute, Kalispell, Montana
  - Premier Research, Trenton, New Jersey
  - Manhattan Medical Research, New York, New York
  - Great Lakes Medical Research, Westfield, New York
  - Metrolina Internal Medicine, P.A., Charlotte, North Carolina
  - Diabetes & Endocrinology Consultants PC, Morehead City, North Carolina
  - Aventiv Research, Columbus, Ohio
  - Intend Research, Norman, Oklahoma
  - IPS Research Company, Oklahoma City, Oklahoma
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Summit Research Network Inc, Portland, Oregon
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Detweiler Family Medicine, Lansdale, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Sudir Bansal M.D. Inc., Warwick, Rhode Island
  - PMG Research of Charleston, LLC, Moncks Corner, South Carolina
  - Chattanooga Research and Medicine (CHARM), Chattanooga, Tennessee
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Southern Endocrinology and Associates PA, Mesquite, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - ClinPoint Trials, LLC, Waxahachie, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Advanced Research Institute, Ogden, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Capital Clincial Research Center, Olympia, Washington
  - Walla Walla Clinic, Walla Walla, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - Prevea Clinic, Inc, Green Bay, Wisconsin
- Argentina (17):
  - Centro Medico CICEMO, Caba, Buenos Aires
  - CEDIC-Centro de Investigaciones Clinicas, Caba, Buenos Aires
  - Investigaciones Medicas IMOBA S.R.L., Caba, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Centro Medico Dr Laura Maffei Investigacion Clinica Aplicada, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Centro de Investigacion y Prevencion Cardiovascular (CIPREC), Ciudad Autonoma de, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - CIPADI, Godoy Cruz, Mendoza Province
  - AXISMED SRL - Bioclinica Research Network, Buenos Aires
  - CENUDIAB, Ciudad Autonoma de Buenos Aire
  - Centro Médico Viamonte, Ciudad Autonoma de Buenos Aire
  - Instituto Centenario, Ciudad Autonoma de Buenos Aire
  - Cemediab - Centro Médico Diabetológico Dr. Alejandro Chertkoff, Ciudad Autonoma de Buenos Aire
  - Mautalen Salud e Investigación - Servicio de Endocrinología, Ciudad Autonoma de Buenos Air
  - Instituto Medico Strusberg, Córdoba
  - Centro Medico Privado San Vicente Diabetes, Córdoba
  - Cent Priva Especiali Médicas Ambulatorias Inve Clin CEMAIC, Córdoba
- Austria (6):
  - Landesklinikum Korneuburg-Stockerau, Standort Stockerau, Stockerau, Lower Austria
  - Universitätsklinikum Graz, Graz, Styria
  - Ordination Dr. Evelyn Fließer-Görzer, Saint Stefan Ob Stainz, Styria
  - VIVIT Institut am LKH Feldkirch, Feldkirch, Vorarlberg
  - KA Rudolfstiftung, Vienna
  - Zentrum für klinische Studien Dr. Ursula Hanusch GmbH, Vienna
- Canada (6):
  - Bailey Clinic, Red Deer, Alberta
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - T. Nemtean Medicine Professional Corporation, Mississauga, Ontario
  - Bluewater Clinical Research Group Inc, Sarnia, Ontario
  - Stayner Medical Clinic, Stayner, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
- Greece (10):
  - Iatriko Palaiou Falirou, Medical Center, Palaió Fáliro, Athens
  - Laiko General Hospital of Athens, Ampelokipoi, Attica
  - Gen Hospital of Athens G Gennimatas, Athens, Attica
  - G.Papanikolaou General Hospital, Eksochi, Thessaloniki
  - Thermi Clinic, Thermi, Thessaloniki
  - Athens Euroclinic, Athens
  - University General Hospital of Larissa, Larissa
  - AHEPA Hospital, Thessaloniki
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
  - Euromedica - General Clinic of Thessaloniki, Thessaloniki
- Hungary (9):
  - Studium Egeszseghaz Kft., Kalocsa, Bács-Kiskun county
  - Kenezy Gyula Korhaz es Rendelointezet, Debrecen, Hajdú-Bihar
  - Grof Esterhazy Korhaz es Rendelointezeti Szakrendelo, Pápa, Veszprém megye
  - Szent Margit Rendelointezet, Budapest
  - ClinDiab Kft., Budapest
  - Strazsahegy Medicina Bt., Budapest
  - TRANTOR 99 Bt., Budapest
  - Kanizsai Dorottya Korhaz, Nagykanizsa
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Israel (9):
  - Maccabi Diabetes Clinic, Grand Canyon, North District, Haifa, Haifa
  - Linn Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Clalit Health Services - Shuali Clinic, Raanana
  - ZIV Medical Center, Safed
  - Sakhnin Community Clinic, Clalit Health Services, Sakhnin
  - Diabetes Medical Center (DMC), Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Azienda Ospedaliera Universitaria Careggi, Florence, Florence
  - Istituto Clinico Humanitas, Rozzano, Milano
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena, SI
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Policlinico Mater Domini, Catanzaro
  - Fondazione Universitaria degli Studi G D'Annunzio, Chieti
  - Ospedale Santa Maria Goretti, Latina
  - Policlinico Giaccone, Palermo
  - Ospedale Civile Maggiore Borgo Trento, Verona
- Mexico (2):
  - Hospital Univ. Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Investigacion en Salud y Metabolismo S.C, Chihuahua City
- Poland (15):
  - NZOZ ZDROWIE Osteo-Medic, Bialystok
  - Poradnia Diabetologiczna SN ZOZ Lege Artis, Bialystok
  - NS ZOZ Osrodek Diabetologiczny " Popula", Bialystok
  - Centrum Badan Klinicznych, PI House, Gdansk
  - NZOZ Salvia s.c., Katowice
  - NZOZ Diab-Endo-Met, Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - Gabinety Terpa, Lublin
  - NZOZ Przychodnia Specjalistyczna MEDICA, Lublin
  - Centrum Medyczne OMEDICA, Poznan
  - Praktyka Lekarska, Poznan
  - Nzoz Neuro - Kard, Poznan
  - NZOZ Przychodnia Specjalistyczna Henryk RudzkiAndrzej Wittek, Ruda Śląska
  - Centralny Szpital Kliniczny MSW, Warsaw
  - Regionalna Poradnia Diabetologiczna, Wroclaw
- Puerto Rico (4):
  - Research and Cardiovascular Corp., Ponce, PR
  - Office: Dr. Luis Rivera Colon, San Juan, PR
  - Clinical Research Puerto Rico, Inc., San Juan
  - GCM Medical Group PSC, San Juan
- Romania (17):
  - S. C. Grandmed S.R.L., Str., Oradea, Bihor County
  - SC Gama Diamed SRL, Mangalia, Constanța County
  - Spitalul Judetean de Urgenta Satu Mare, Satu Mare, Jud Satu-Mare
  - CMI DNBM Dr. Pop Lavinia, Baia Mare, Maramureş
  - Cosamext SRL, Târgu Mureş, Mureș County
  - SC Diabmed Dr Popescu Alexandrina SRL, Ploieşti, Prahova
  - SC Dianutrilife Medica SRL, Ploieşti, Prahova
  - Centrul Medical Dr. Negrisanu, Timișoara, Timiș County
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed SRL, Brasov
  - Cabinetul Medical Nicodiab SRL, Bucharest
  - Easydiet SRL, Bucharest
  - SC Nutrilife SRL, Bucharest
  - SC Medcon SRL, Buzău
  - Centrul Medical Unirea SRL, Cluj-Napoca
  - Cabinet Medical Urodiamed S.R.L., Craiova
  - Milena Sante SRL, Galati
  - SC Olimpia Med SRL, Iași
- Russia (6):
  - Regional Clinical Hospital, Saratov, Russian Federation
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Arkhangelsk the first city clinical hospital, Arkhangelsk
  - Rostov State Medical University, Rostov-on-Don
  - City Hospital of Saint Martyr Elizabeth, Saint Petersburg
  - SPb GUZ "Diagnostic Center #85", Saint Petersburg
- Slovakia (9):
  - Human care s.r.o., Košice, Slovak Republic
  - MediVet s.r.o., Malacky, Slovak Republic
  - Areteus s.r.o., Trebišov, Slovak Republic
  - Diacrin s.r.o., Bratislava
  - Noemis, s.r.o., Nové Mesto nad Váhom
  - FUNKYSTUFF s.r.o., Nové Zámky
  - MUDr. Jan Culak, s.r.o., Prievidza
  - DIA-MED CENTRUM s.r.o., Púchov
  - Tatratrial s.r.o., Rožňava
- Spain (14):
  - Hospital Infanta Luisa, Seville, Andalusia
  - Clinica Juaneda, Palma de Mallorca, Balearic Islands
  - Corporació Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques De Valdecilla, Santander, Cantabria
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Instituto de Ciencias medicas, Alicante
  - Clinica San Pedro, Almería
  - Centre Medico Teknon, Barcelona
  - Hospital Clinico Universitario San Cecilio, Granada
  - Virgen de Las Nieves, Granada
  - Centro Especialidades San Jose Obrero (Barbarela), Málaga
  - Clinica Nuevas Tecnologias en Diabetes y Endocrinologia, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Policlinica Galileo, Teruel
- Taiwan (3):
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi-Mei Medical Center, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Ferdinand KC, Dunn J, Nicolay C, Sam F, Blue EK, Wang H. Weight-dependent and weight-independent effects of dulaglutide on blood pressure in patients with type 2 diabetes. Cardiovasc Diabetol. 2023 Mar 9;22(1):49. doi: 10.1186/s12933-023-01775-x. PMID 36894938
- [Derived] Cox DA, Wang H, Nicolay C, Bethel MA. Effect of expanded dulaglutide weekly doses (3.0 mg and 4.5 mg) on cardiovascular disease risk factors in participants with type 2 diabetes at increased cardiovascular disease risk: a post hoc analysis of the AWARD-11 study. Diabetes Obes Metab. 2022 Sep;24(9):1770-1778. doi: 10.1111/dom.14762. Epub 2022 May 29. PMID 35546790
- [Derived] Frias JP, Bonora E, Nevarez Ruiz L, Li YG, Yu Z, Milicevic Z, Malik R, Bethel MA, Cox DA. Efficacy and Safety of Dulaglutide 3.0 mg and 4.5 mg Versus Dulaglutide 1.5 mg in Metformin-Treated Patients With Type 2 Diabetes in a Randomized Controlled Trial (AWARD-11). Diabetes Care. 2021 Mar;44(3):765-773. doi: 10.2337/dc20-1473. Epub 2021 Jan 4. PMID 33397768
- See also: A Study of the Efficacy and Safety of Dulaglutide (LY2189265) in Participants With Type 2 Diabetes (AWARD-11) — https://www.lillytrialguide.com/en-US/studies/adult-type-2-diabetes/GBGL#?postal=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg
Started | 612 | 616 | 614
Received at Least One Dose of Study Drug | 612 | 616 | 614
Completed | 556 | 549 | 560
Not Completed | 56 | 67 | 54
Not completed — Adverse Event | 5 | 7 | 10
Not completed — Death | 3 | 4 | 4
Not completed — Lost to Follow-up | 15 | 16 | 17
Not completed — Physician Decision | 2 | 0 | 2
Not completed — Withdrawal by Subject | 25 | 36 | 18
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Site Closure | 3 | 1 | 2
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Participant Duplicated at Another Site | 0 | 0 | 1
Not completed — Primary Care Physician Recommendation | 0 | 1 | 0
Not completed — Relocated to Another Country | 0 | 1 | 0
Not completed — Participant was in Rehabilitation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg | Total
Number analyzed (Participants) | 612 | 616 | 614 | 1842
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.7) | 56.9 (10.2) | 56.6 (10.2) | 57.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 288 | 296 | 898
  Male | 298 | 328 | 318 | 944
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 214 | 214 | 213 | 641
  Not Hispanic or Latino | 369 | 363 | 371 | 1103
  Unknown or Not Reported | 29 | 39 | 30 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 30 | 26 | 32 | 88
  Asian | 13 | 18 | 14 | 45
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 3 | 5
  Black or African American | 28 | 31 | 23 | 82
  White | 529 | 521 | 530 | 1580
  More than one race | 11 | 19 | 12 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 96 | 97 | 97 | 290
  Romania | 77 | 78 | 78 | 233
  Hungary | 25 | 24 | 24 | 73
  United States | 169 | 169 | 170 | 508
  Russia | 9 | 10 | 10 | 29
  Spain | 19 | 20 | 19 | 58
  Greece | 33 | 34 | 33 | 100
  Canada | 12 | 11 | 12 | 35
  Austria | 4 | 4 | 5 | 13
  Taiwan | 5 | 5 | 5 | 15
  Poland | 56 | 56 | 55 | 167
  Mexico | 37 | 38 | 36 | 111
  Italy | 9 | 8 | 8 | 25
  Slovakia | 43 | 44 | 44 | 131
  Israel | 18 | 18 | 18 | 54
Hemoglobin A1C (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.64 (0.94) | 8.63 (1.00) | 8.64 (0.91) | 8.64 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c) From Baseline
Description: HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. The Least Squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included the independent variables:Baseline + Pooled Country + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 36
Population: All participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline HbA1c value, excluding data post treatment discontinuation and/or initiation of new antihyperglycemic medications.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg
Number analyzed (Participants) | 523 | 521 | 526
Percentage of HbA1c | -1.53 (0.04) | -1.71 (0.04) | -1.87 (0.04)
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 3 mg; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.29 to -0.06]
Statistical Analysis 2: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 4.5 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.45 to -0.22]

2. Secondary Outcome: Change in Body Weight From Baseline
Description: Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with independent variables: Baseline + Baseline HbA1c group + Pooled Country + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 36
Population: All participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline body weight value, excluding data post treatment discontinuation and/or initiation of new antihyperglycemic medications.
Measure: Least Squares Mean (Standard Deviation); unit: Kilograms (Kg)
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg
Number analyzed (Participants) | 522 | 520 | 526
Kilograms (Kg) | -3.1 (0.19) | -4.0 (0.19) | -4.7 (0.19)
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 3 mg; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.9, 95% CI 2-sided [-1.4 to -0.4]
Statistical Analysis 2: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 4.5 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.6, 95% CI 2-sided [-2.1 to -1.1]

3. Secondary Outcome: Percentage of Participants Achieving HbA1c Target <7.0%
Description: Percentage of participants achieving HbA1c target <7.0%.
Time Frame: Week 36
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg
Number analyzed (Participants) | 523 | 521 | 526
percentage of participants | 56.98 | 64.68 | 71.48
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 3 mg; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.12 to 1.98]
Statistical Analysis 2: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 4.5 mg; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.65 to 3.01]

4. Secondary Outcome: Change in Fasting Serum Glucose (FSG) From Baseline
Description: Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with covariates: Baseline + Baseline HbA1c group + Pooled Country + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 36
Population: All participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline FSG value, excluding data post treatment discontinuation and/or initiation of new antihyperglycemic medications.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg
Number analyzed (Participants) | 510 | 509 | 514
milligrams per deciliter (mg/dL) | -44.2 (1.50) | -47.9 (1.50) | -52.3 (1.50)
Statistical Analysis 1: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 3 mg; Test type: Superiority; p = 0.084, Mixed Models Analysis; Mean Difference (Net) = -3.7, 95% CI 2-sided [-7.8 to 0.5]
Statistical Analysis 2: Comparison: Dulaglutide 1.5 mg vs Dulaglutide 4.5 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -8.1, 95% CI 2-sided [-12.3 to -3.9]

5. Secondary Outcome: Rate of Documented Symptomatic Hypoglycemic Episodes
Description: Hypoglycemia was defined as blood glucose < 54 mg/dL, excluding post-rescue records. Estimate is based on Group Mean from negative binomial model. The negative binomial model for post-baseline comparisons between treatments and control group: Number of episodes = Pooled Country + HbA1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Week 36
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Error); unit: Episodes/participant/365.25 days
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg
Number analyzed (Participants) | 612 | 616 | 614
Episodes/participant/365.25 days | 0.02 (0.01) | 0.00 (0.00) | 0.02 (0.01)

6. Secondary Outcome: Pharmacokinetic (PK): Steady-state Maximum Concentration(Cmax,ss)
Description: Pharmacokinetic (PK): Steady-state Maximum Concentration(Cmax,ss).
Time Frame: Week 4, Week 12, Week 36, Week 52
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (90% Confidence Interval); unit: nanogram/milliliter (ng/mL)
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg
Number analyzed (Participants) | 612 | 616 | 614
nanogram/milliliter (ng/mL) | 79.6 [77.7 to 81.7] | 159 [155 to 163] | 238 [232 to 243]

7. Secondary Outcome: Pharmacokinetic (PK): Area Under the Curve AUC (0-168)ss at Steady State
Description: Pharmacokinetic (PK): Area Under the Curve AUC (0-168)ss at Steady State.
Time Frame: Week 4, Week 12, Week 36, Week 52
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (90% Confidence Interval); unit: nanogram*hour/milliliter (ng*h/mL)
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg
Number analyzed (Participants) | 612 | 616 | 614
nanogram*hour/milliliter (ng*h/mL) | 11200 [10900 to 11500] | 22300 [21800 to 22900] | 33400 [32700 to 34200]

ADVERSE EVENTS:
Time Frame: Up to Week 56
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Dulaglutide 1.5 mg | Dulaglutide 3 mg | Dulaglutide 4.5 mg
All-Cause Mortality (participants affected / at risk) | 3/612 | 4/616 | 4/614
Serious Adverse Events (participants affected / at risk) | 53/612 | 45/616 | 38/614
Other Adverse Events (participants affected / at risk) | 156/612 | 190/616 | 195/614
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dulaglutide 1.5 mg (N=612) | Dulaglutide 3 mg (N=616) | Dulaglutide 4.5 mg (N=614)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Medical device site joint inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Perinephric abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
West nile viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ecg signs of myocardial ischaemia (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram t wave inversion (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Plica syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/314 (1) | 0/288 (0) | 0/296 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/298 (1) | 0/328 (0) | 0/318 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/314 (1) | 0/288 (0) | 0/296 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic mononeuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Wernicke's encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/314 (0) | 2/288 (2) | 0/296 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0/314 (0) | 1/288 (1) | 0/296 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/314 (0) | 0/288 (0) | 1/296 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dulaglutide 1.5 mg (N=612) | Dulaglutide 3 mg (N=616) | Dulaglutide 4.5 mg (N=614)
Diarrhoea (Gastrointestinal disorders) | 48 (83) | 75 (118) | 70 (176)
Dyspepsia (Gastrointestinal disorders) | 17 (26) | 33 (56) | 18 (35)
Nausea (Gastrointestinal disorders) | 87 (121) | 99 (180) | 106 (192)
Vomiting (Gastrointestinal disorders) | 40 (63) | 57 (89) | 64 (108)
Nasopharyngitis (Infections and infestations) | 29 (38) | 33 (41) | 39 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT03495102/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT03495102/SAP_001.pdf